CLINICAL TRIAL: NCT06121960
Title: Evaluation of Respiratory Function During Self-induced Cognitive Trance
Acronym: SPIROTRANSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHMS22009
Record Dates: First submitted 2023-05-26; First posted 2023-11-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Function
Keywords: spirometry; TCAI (Cognitive-induced trance)
MeSH Terms: conditions — Respiratory Aspiration | interventions — Spirometry

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, non-randomized, open-label study.
Masking Description: Person with expertise in the practice of TCAI. (at least 6 months, in order to be able to control the depth of the trance and to have a motor control allowing the realization of a spirometry)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventionnal (Experimental): Measure DEP, DEM25, DEM 50, DEM 75, FVC, Inspiratory capacity, SpO2, Respiratory rate before, during, or after the state of self-induced cognitive trance Evolution of the feeling of self-efficacy, assessed by questionnaire.
  Interventions: Diagnostic Test: spirometry

INTERVENTIONS:
Diagnostic Test: spirometry — Inclusion visit:
  Performing spirometry.
  Visit 2 (in the month following the inclusion visit):
  Induction of a self-induced cognitive trance by the participant; performance of spirometry before, during the trance then 8 minutes after the end of the trance Actimetry during trance

SUMMARY:
The goal of this Prospective, monocentric, non-randomized, open-label study aimed at evaluating the variation of FEV1 during a state of self-induced cognitive trance participant population: Person with expertise in the practice of TCAI can be inclued. (at least 6 months, in order to be able to control the depth of the trance and to have a motor control allowing the realization of a spirometry)

The main question:

Study the significant variation of FEV1 before, during, or after the state of self-induced cognitive trance

DETAILED DESCRIPTION:
Primary objective : Study the significant variation of FEV1 before, during, or after the state of self-induced cognitive trance judgment criteria:

Significant variations in:

PEF PEF25 PEF50 PEF75 FVC Inspiratory capacity, SpO2 Respiratory rate before, during, or after the self-induced cognitive trance state Evolution of the feeling of self-efficacy, assessed by questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Person over 18 years old
* Person with expertise in the practice of TCAI. (at least 6 months, in order to be able to control the depth of the trance and to have a motor control allowing the realization of a spirometry)
* Person affiliated with social security or beneficiary of such a scheme.
* Person having given, in writing, their free and informed consent to participate in the study

Exclusion Criteria:

* Person deprived of liberty by judicial or administrative decision, person subject to a measure of legal protection.
* Exclusion period for other studies
* Person likely, according to the investigator's assessment, not to be cooperative or respectful of the obligations inherent in participation in the study
* Person with a psychiatric, neurological or cardiovascular disease.
* Person with a chronic respiratory disease, for example: asthma, COPD, interstitial lung disease, bronchial dilation, cystic fibrosis,
* Person with a history of exercise-induced bronchospasm.
* Person taking inhaled treatments (corticotherapy, bronchodilators, anticholinergics)
* Pregnant woman (declarative).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
FEV during a state of self-induced cognitive trance | 3 month
  variation of forced exhaled volume in one second between pre and post phase of cognitive transe

SECONDARY OUTCOMES:
PEF during a state of self-induced cognitive trance | 3 month
  variation of PEF between pre, per and post phase of cognitive transe
DEM25/50/75 during a state of self-induced cognitive trance | 3 month
  variation of DEM25/50/75 between pre, per and post phase of cognitive transe
inspiratory capacity during a state of self-induced cognitive trance | 3 month
  variation of inspiratory capacity between pre, per and post phase of cognitive transe
respiratory rate during a state of self-induced cognitive trance | 3 month
  variation of respiratory rate between pre, per and post phase of cognitive transe
SpO2 during a state of self-induced cognitive trance | 3 month
  variation of SpO2 between pre, per and post phase of cognitive transe
FVC during a state of self-induced cognitive trance | 3 month
  variation of FVC between pre, per and post phase of cognitive transe

CONTACTS AND LOCATIONS:
Overall Officials: Pierre IDEE, Study Director — CH Metropole Savoie
Locations (1):
- Centre Hospitalier Metropole Savoie, Chambéry, Savoie, France

IPD SHARING:
Plan to Share IPD: No